CLINICAL TRIAL: NCT05368324
Title: Improvement of Planning Skills in Daily Life in Children and Adolescents With ADHD Through a Virtual Reality System: CogFun-RV
Brief Title: Improvement of Planning Skills in Children and Adolescents With ADHD Through a Virtual Reality System: CogFun-RV
Acronym: CogFun-RV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Dulce Romero Ayuso, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: UGranadaII
Record Dates: First submitted 2022-05-01; First posted 2022-05-10 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, with a control group on the waiting list.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All participants will be evaluated by an independent evaluator who will be blinded. The statistician will also be blinded, will not participate in the evaluation or intervention. For analysis it will only be revealed as group A or group B. Only when the analyzes have been completed will the exact nature of the groups be revealed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CogFun-RV (Experimental): It consists of 12 sessions, each lasting 75 minutes for each children. Parallel parents will participate in the parental guidance and psychoeducation program with one of the two therapists assigned to the child.
  Interventions: Behavioral: CogFun-RV
- Control group on waiting list (Other): After 6 months, the participants of the control group on the waiting list will be invited to participate if the results of the analysis show positive effects of the intervention.
  Interventions: Behavioral: CogFun-RV

INTERVENTIONS:
Behavioral: CogFun-RV — CogFun-RV intervention combines training in daily living skills, organization, task planning, time organization, emotional regulation, self-esteem and mindfulness in children and the parents. It consists of 12 sessions, each lasting 75 minutes. Parents will participate in the parental guidance and psychoeducation program with one of the two therapists assigned to the child. As it is a program of a simultaneous nature, excessive impact on the daily life of families is avoided. All sessions will be carried out individually.

SUMMARY:
The main aim is to know the effectiveness of a program, CogFun-VR, through the use of immersive virtual reality, to improve executive skills, such as self-regulation, organization, planning and time management in life. of children and adolescents with ADHD, between 9 and 16 years old.

The study design is a randomized clinical trial, with a control group on a waiting list. The estimated sample size is 82 participants: 41 in the experimental group and 41 in the control group.

Participants will be randomly assigned to one of the two groups. Four measurements of the variables of interest will be conducted, in the beginning, after the 12-week duration of the intervention, at 3 months and 6 months as a follow-up. The BRIEF, SNAP-IV, SDQ, EQi: YV and several subtests of the WISC-%, BADS and NEPSY-II will be used. All participants will be assessed by an independent evaluator who will be blinded. The intervention program is manualized to assess its integrity and reliability.

DETAILED DESCRIPTION:
Planning skills are one of the difficulties that children with ADHD show, being reflected in four of the nine symptoms of inattention according to the DSM-5. In addition, these skills have been associated with performance in different daily, academic, work and leisure activities.

The main objective of the study is to know the effectiveness of an innovative treatment to improve executive skills, such as planning, organization and time management in daily life in children and adolescents between 9 and 16 years old with a diagnosis of ADHD, through a program multimodal of 12 individual sessions of 75 minutes.

The study design is a randomized clinical trial, with a control group on a waiting list. The estimated number of participants is 82, 41 participants in the experimental group and 41 children in the control group on the waiting list. Participants will be randomly assigned to one of two groups. Three measurements of the variables of interest will be made. All participants will be evaluated by an independent evaluator who will be blinded. The intervention program is manualized in order to assess its integrity and reliability. All sessions are divided into two parts: 1) intervention through an immersive virtual reality system, called COGFUN-RV, lasting 30 minutes and 2) teaching strategies to improve cognitive and emotional self-regulation skills. for another 30 minutes. Each session will include practice, at home or at school, of the strategies learned until the next session. The intervention proposal incorporates 15 minutes of psychoeducation with the parents in each session. The project has been submitted for approval to the Ethics and Human Research Committee of the University of Granada, as well as to the PEIBA. All legal guardians will have to give their informed consent and authorization to participate in the project.

The program represents a novelty in the current treatment for several reasons. First, until now most programs have focused only on basic executive functions, such as working memory, inhibitory control, or cognitive flexibility. Instead, this proposal focuses especially on advanced executive functions, such as planning, organization, time management, and problem solving. Secondly, the main approach is through a virtual reality system, in which the child must plan, manage time, organize the action and regulate its emotions, according to the different actions carried out in the activity. The main characteristic of the virtual proposal is to increase the transfer to daily life and, therefore, the ecological validity.

ELIGIBILITY:
Inclusion criteria:

* Age between 9 and 17 years
* Clinical diagnosis of ADHD
* With stable pharmacological treatment

Exclusion criteria:

* Children with disorders comorbid with ASD and severe behavioural disorders
* With other non-pharmacological treatments
* That they start a new pharmacological or non-pharmacological treatment during the duration of the study (they will not be considered for the analysis of the results).
* Have visual deficits that prevent the use of virtual reality glasses
* Present symptoms of Cybersickness

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
Weiss Functional Impairment Rating Scale-Parent Form for assessing ADHD | After the Intervention (12 weeks)
  The Weiss Functional Impairment Rating Scale- Parent Form (WFIRS-P) is a 50-item scale that assesses functional impairment on six clinically relevant domains typically affected in attention-deficit/hyperactivity disorder (ADHD)
Weiss Functional Impairment Rating Scale-Parent Form for assessing ADHD | At 3 months
  The Weiss Functional Impairment Rating Scale Parent Form (WFIRS-P) is a 50-item scale that assesses functional impairment on six clinically relevant domains typically affected in attention-deficit/hyperactivity disorder (ADHD)
Weiss Functional Impairment Rating Scale-Parent Form for assessing ADHD | At 6 months
  The Weiss Functional Impairment Rating Scale- Parent Form (WFIRS-P) is a 50-item scale that assesses functional impairment on six clinically relevant domains typically affected in attention-deficit/hyperactivity disorder (ADHD)
Self-assessment of daily time management in children (TIME-S) | After the intervention: 12 weeks
  Self-assessment for children with disabilities ages 10-17 ability of time perception, time orientation andknowledge on time management in children 10-17 years old
Self-assessment of daily time management in children (TIME-S) | At 3 months
  Self-assessment for children with disabilities ages 10-17 ability of time perception, time orientation andknowledge on time management in children 10-17 years old
Self-assessment of daily time management in children (TIME-S) | At 6 months
  Self-assessment for children with disabilities ages 10-17 ability of time perception, time orientation andknowledge on time management in children 10-17 years old

SECONDARY OUTCOMES:
Assessment of Executive Function and Sensory Processing (EPYFEI) | Before and after the intervention (12 weeks)
  Questionnaire for parent.Scores above 46.5 points indicate that there is a deficit in executive functioning in daily life. The higher the score, the worse the result.
Conners Behavior Questionnaire for Parents (SNAP-IV) | Before and after the intervention (12 weeks)
  Behavior scale for children and adolescents with ADHD. Higher score mean worse outcome.
Zoo Map Subtest | Before and after the intervention (12 weeks)
  Planning Skills Cognitive Test.The number of errors is scored, the higher the score, the worse the results. The scores are between 0 and 10.
Stroop Test | Before and after the intervention (12 weeks)
  Cognitive test of selective attention and interference inhibition.The score can be positive or negative. If the score is negative, below zero, it indicates that there are difficulties in inhibiting interference from the environment.
Trail Making Test | Before and after the intervention (12 weeks)
  Cognitive test of sustained and alternating attention.The number of errors and the time it takes to complete the task are collected. Scores vary by age. The higher the number of errors and the longer the execution time, the worse the attention.
Digit test | Before and after the intervention (12 weeks)
  Attentional Span and Working Memory.The higher the score, the better the results. Normal scores range between 6 and 9 digits of attention span.
Emotional intelligence scale EQ-i:Yv | Before and after the intervention (12 weeks)
  Emotional intelligence scale for children and young people.The higher the score, the better the results. The average scores are between 90-100 points.
Strengths and Difficulties Questionnaire (SDQ)-parents | Before and after the intervention (12 weeks)
  Assessment of behavioural problems.The minimum score is 0 and the maximum is 40. The normal score is between 0-13 points. A score greater than 17 was considered abnormal.

IPD SHARING:
Plan to Share IPD: No